## **ClinicalTrials.gov-Compliant Summary**

Study Title: Hand Joints Hypermobility and Its Relation to Muscular Strength Among Physical Therapy Students: A Cross-Sectional Study

Brief Summary: This observational cross-sectional study aims to assess the prevalence of hand joint hypermobility among first-year physical therapy students and examine the correlation between hypermobility severity and muscular strength. The study will involve standardized assessments of finger joint hyperextension and grip strength.

Study Type: Observational | Model: Cross-Sectional | Time Perspective: Prospective

Study Population: First-year physical therapy students enrolled at Horus University, Egypt.

Estimated Enrollment: 400 participants

Eligibility Criteria: Inclusion: First-year physical therapy students (academic year 2023/2024), Age 18–20 years, No previously diagnosed systemic conditions associated with hypermobility. Exclusion: Students enrolled in any other academic year, Failure to attend in-person assessment, Age outside 18–20 years.

Age Range: 18-20 years | Sex: Male and Female

Outcome Measures: Primary: Degree of hand joint hypermobility assessed using a universal goniometer. Secondary: Grip strength measured using a handheld dynamometer.

Study Location: Faculty of Physical Therapy, Horus University, Egypt

Principal Investigator: Dr. Ehab Ali Abdallah | Email: Eabdallah@horus.edu.eg

Ethics Approval: Approved by Faculty of Physical Therapy Research Ethics Committee.

Potential Benefits: Early identification of hypermobility may improve clinical performance and guide preventive interventions for physical therapy students.

Document Date: 2022-11-09